CLINICAL TRIAL: NCT07400497
Title: Family Foundations for Special Education
Brief Title: Family Foundations for Special Education Trial
Acronym: SS-SE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Public Health Management Corporation (Other); William Penn Foundation (Other)
Responsible Party: Principal Investigator, Mark Feinberg, Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00025916; 218-23 (Other Grant/Funding Number: William Penn Foundation)
Record Dates: First submitted 2026-01-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mental Health
Keywords: parenting education; children with disabilities; children with challenging behaviors; parenting relationships; Coparenting; Special Education
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive FF-SE in six virtual learning sessions to receive information on the special education system and methods to improve communications and working together as co-parents to enhance their IEP experience. The duration of each session will be between 1 to 1 ½ hour long and will be scheduled weekly according to the participants preferred scheduled. A workbook with supporting documents for each session will be mailed and/or emailed to each participant prior to the start of the sessions.
  Interventions: Behavioral: Family Foundations for Special Education
- Group B (No Intervention): Group B will have access to existing standard supports available to families entering the special education system.

INTERVENTIONS:
Behavioral: Family Foundations for Special Education — Families in the intervention group receive the new enhanced supports and participate in six private virtual learning sessions focused on understanding the special education system, improving communication, and enhancing collaboration as co-parents in the IEP process. Each session lasts 60-90 minutes and will be scheduled weekly according to the participants preferred schedule, including evenings and weekends. A workbook with supporting documents for each session will be sent to each participant prior to the start of the sessions.
  Other Names: FF-SE
  Arms: Group A

SUMMARY:
The goal of this clinical trial is to assess the program's impact on parent self-efficacy and co-parental support around (a) accessing health and educational services and (b) parenting for co-parents of children with disabilities entering the Special Education system before their first Individualized Education Program (IEP) meeting. The main questions it aims to answer are: Does the program improve co-parenting support and coordination and parent efficacy in accessing services for and parenting their child? Does the program improve parent mental health, service access, engagement, and adherence? Does the program improve parenting quality? Does the program improve child adjustment (mental and behavioral health, academic engagement)? Researchers will compare pretest and posttest questionnaires from Treatment Group A with Control Group B to see if the program improves parent and child well-being, co-parenting relations, relations with service providers, ability to access services and meaningfully participate in IEP and other meetings.

Participants will:

* Complete pre- and post-test questionnaires
* Treatment Group A will participate in 6 learning sessions, each 1 hour to 1½ hour long, over a 6-8 week period

ELIGIBILITY:
Inclusion Criteria:

* Parents/parental figures who are over the age of 18, and are involved in childrearing together.
* Coparenting a child being evaluated for special education services
* Has not yet had their first IEP meeting.
* The target child must attend a Philadelphia elementary school (K-8).
* The target child must be the first child in the family to go through the IEP process.
* Co-parents must be fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Coparenting Relationship Questionnaire | From enrollment to the last learning session for intervention group, approximately 2 months after enrollment for the control group.
  A validated, parent-report questionnaire on key dimensions of the coparenting relationship.
Parenting Sense of Competence Scale | From pretest to two months post-intervention
  Parent-reported, 17 item scale (Gibaud-Wallston & Wandersman, 1978) assessing parent self-efficacy in accessing services for their child. Higher scores reflect higher degree of sense of competence.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No